CLINICAL TRIAL: NCT03958318
Title: The Effectiveness of a Multi-component Exercise Program Plus Oral Nutritional Supplementation, on the Functional Capacity in Frail Institutionalized Older Adults.
Brief Title: Multi-component Exercise Program and Nutritional Supplementation in Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: University CEU-UCH
Record Dates: First submitted 2019-01-10; First posted 2019-05-22 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Fragility
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Multi-modal exercise program
  Interventions: Other: Exercise
- Exercise plus nutritional suplementation (Experimental): Multi-modal exercise program plus nutritional suplementation
  Interventions: Other: Exercise plus nutritional suplementation
- Control (No Intervention): No interventions

INTERVENTIONS:
Other: Exercise plus nutritional suplementation — For 6 months, all participants in the exercise plus nutritional supplementation group will be performing a three-week non-consecutive exercises programme at the facility. All exercises will be undertaken in a large indoor room. The exercise routine will be based on the Otago exercise programme.
  Arms: Exercise plus nutritional suplementation
Other: Exercise — For 6 months, all participants in the exercise group will be performing a three-week non-consecutive exercises programme at the facility. All exercises will be undertaken in a large indoor room. The exercise routine will be based on the Otago exercise programme.
  Arms: Exercise

SUMMARY:
The objective of this study is to evaluate the effects of a multi-modal group-based exercise program and nutritional supplementation on physical performance in frail institutionalized older adults.

Participants will be randomly allocated to the intervention groups; exercise (EG) or exercise plus nutritional supplementation (SG), or to the control group (CG). During 6 months, participants in the intervention groups will be performing the exercise routine based on the Otago exercise programme. Additionally, participants in the SG will receive a daily oral nutritional supplement.

DETAILED DESCRIPTION:
Objectives: Evaluate the effects of a multi-modal group-based exercise program and nutritional supplementation on physical performance and the capacity to perform daily tasks in frail institutionalized older adults.

Design: Randomized controlled trial, with a 6-month intervention period. Participants: 122 frail institutionalized older adults aged 65 and older with no cognitive impairment.

Intervention: After a baseline assessment, the participants will be randomly assigned to the control group or one of two intervention groups; multi-modal exercise program (EG) or exercise plus nutritional supplementation (SG). During 6 months, participants in the intervention groups will be performing the exercise routine based on the Otago exercise programme. Additionally, participants in the SG will receive a daily oral nutritional supplement.

Measurements: The primary outcome measure will be mobility measured with the timed up and go test. Secondary outcomes will be the functional balance, hand-grip strength, lower limb functional capacity, gait speed and distance covered during the 6-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years;
* Frail institutionalized.

Exclusion Criteria:

* Cognitive impairment;
* Fracture;
* Neurological disorder;
* Unable to follow verbal instructions;
* Score lower than 60 in the Barthel Index.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 5-10 minutes
  The participants will be instructed to stand up from a standard chair of 45 cm height, walk 3 metre, turn around a cone, return to the chair, and sit down again in the shortest time possible without running. Two trials will be performed, and the quicker time in seconds will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Vicent Benavent Caballer, Alfara del Patriarca, Spain

REFERENCES:
- [Derived] Garcia-Gollarte F, Mora-Concepcion A, Pinazo-Hernandis S, Segura-Orti E, Amer-Cuenca JJ, Arguisuelas-Martinez MD, Lison JF, Benavent-Caballer V. Effectiveness of a Supervised Group-Based Otago Exercise Program on Functional Performance in Frail Institutionalized Older Adults: A Multicenter Randomized Controlled Trial. J Geriatr Phys Ther. 2023 Jan-Mar 01;46(1):15-25. doi: 10.1519/JPT.0000000000000326. Epub 2021 Aug 19. PMID 34417416